CLINICAL TRIAL: NCT04408248
Title: AKI Biomarkers for Prediction of Acute Kidney Injury in Critically Ill Patients With COVID-19 and Respiratory Disease
Brief Title: AKI Biomarkers in Coronavirus(COVID)-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: University Hospital Muenster (Other)
Responsible Party: Sponsor
Other Study IDs: 283675
Record Dates: First submitted 2020-05-27; First posted 2020-05-29 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: COVID; Acute Respiratory Failure; Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The investigators will collect blood and urine samples for biomarker measurement at the following time points: at the time point of study inclusion, 12h, 24h, 36h, 48h, 60h, and 72h after inclusion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19 patients with acute respiratory disease: Adult patients with COVID-19 and moderate or severe respiratory disease

SUMMARY:
This research aims to investigate the role of daily measurement of urinary cell cycle arrest markers and other serum and urinary biomarkers to predict the development of acute kidney injury in critically ill patients with COVID-19 and acute respiratory disease.

DETAILED DESCRIPTION:
COVID-19 is a rapidly evolving pandemic with approximately 5% of all patients requiring admission to an intensive care unit. In critically ill patients with COVID-19, acute respiratory disease and acute kidney injury (AKI) are very common. Patients with AKI have an increased risk of mortality, especially renal replacement therapy (RRT) is required. The latest Intensive Care National Audit & Research Centre (ICNARC) report shows a 77% ICU mortality in patients with COVID-19 who require mechanical ventilation and RRT.

COVID-19 associated AKI is still poorly understood. The exact underlying pathophysiology remains unknown. Furthermore, there are no specific strategies to prevent or treat AKI. Management is supportive consisting of fluid and haemodynamic optimization, discontinuation of nephrotoxic drugs and prevention of nephrotoxic exposures. Ideally, AKI needs to be recognized as early as possible for these supportive measures to be effective.

Early prediction of AKI may be valuable to optimize management and improve outcomes. In critically ill patients without COVID-19, the two cell-cycle arrest markers, tissue inhibitor of metalloproteinases-2 (TIMP-2) and insulin-like growth-factor binding protein 7 (IGFBP7), have been shown to predict the development of AKI. Whether these new biomarkers also predict the development of AKI in critically ill patients with COVID-19 is unknown.

The aim of this project is to explore whether urinary cell cycle arrest markers and other renal biomarkers have a role in predicting AKI in critically ill patients with COVID-19 and acute respiratory disease. The results will advance the understanding of this disease and serve to develop strategies for individualized management of this high-risk group.

ELIGIBILITY:
Inclusion Criteria:

1. Moderate or severe respiratory disease as defined by Berlin criteria
2. COVID-19 positive
3. Age ≥ 18 years

Exclusion Criteria:

1. pre-existing AKI
2. severe chronic kidney disease (CKD) with estimated glomerular filtration rate (eGFR) <20ml/min
3. end-stage renal failure on regular dialysis
4. kidney transplant within the last 12 months
5. pregnancy
6. breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COVID-19 patients with moderate or severe respiratory disease
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-08-20 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Any stage of acute kidney injury | 7 days
  As defined by Kidney Diseases: Improving Global Outcome

SECONDARY OUTCOMES:
need for RRT in first 7 days | 7 days
  Renal replacement therapy requirement at the clinicians' discretion
Mortality | 7 and 28 days
  ICU mortality
Duration of mechanical ventilation | 7 and 28 days
  Duration
Duration of vasopressor support | 7 and 28 days
  Duration

CONTACTS AND LOCATIONS:
Overall Officials: Marlies Ostermann, MD, PhD, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust
Locations (1):
- Guy's & St Thomas' Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided